CLINICAL TRIAL: NCT03735641
Title: Evaluation of the Postoperative Effect of Expanded Pedicled Deltopectoral Flap to Repair the Facial-Cervical Scars
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20182035-C-1
Record Dates: First submitted 2018-10-17; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-09

CONDITIONS: Surgical Flaps; Skin Pigmentation; Sensory Defect
Keywords: Expanded Pedicled Deltopectoral Flap; skin color; Sensory recovery
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- postoperative: Expanded Pedicled Deltopectoral Flap is a type of surgical flap that has been cut away from surrounding areas for transplantation.The postoperative patients are studied . Tested sensory recovery,skin color and Skin elasticity
  Interventions: Procedure: Expanded Pedicled Deltopectoral Flap

INTERVENTIONS:
Procedure: Expanded Pedicled Deltopectoral Flap — Expanded Pedicled Deltopectoral Flap is a type of surgical flap

SUMMARY:
This study evaluates the effect of Expanded Pedicled Deltopectoral Flap on facial-cervical scars repair, including flap sensation, L*a*b* value,flap's elasticity,melanin content, hemoglobin content, and evaluation of scar and patient, doctor, and third-party satisfaction

DETAILED DESCRIPTION:
The scars of face and neck caused by burning often show as large faciocervical scar.Important areas of current focus in face and neck scars management are functional outcomes and quality of patient life.The deltopectoral flap was first described by Bakamjian in 1965, and was recognized as one of the first choices for facial reconstruction, as the texture, color of the flap skin is similar to the facial skin. Since the tissue expansion technique was used to the flap, the flap became one of the best choices for the facial defect reconstruction,especially for Asian patients. It can be used with pedicled or free transferred.Complications at the donor or recipient site have been widely reported and often include dilator exposure,the flap blood circulation disorder and delayed healing, but the pattern of sensory recovery ,flap's elasticitycolor change have been studied less well.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent Expanded Pedicled Deltopectoral Flap to repair facial-cervical scars in 2006 -2018.
2. In compliance with ethical requirements, patients were voluntarily tested and signed informed consent.

Exclusion Criteria:

1. Peripheral neuropathy
2. Serious aphasia or cognitive impairment, and first-degree relatives can not get in touch.
3. Can not follow up
4. Allergic constitution
5. Connective tissue disease
6. Hormone or chemotherapy drugs are being used.
7. Diabetes

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who underwent Expanded Pedicled Deltopectoral Flap to repair facial-cervical scars in 2006 -2018
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Flap Color（the value of L*a*b*） | 3 month later
  The Antera 3D is a camera for image acquisition and analysis of the skin.Every color is expressed in a three-dimensional coordinate system in terms of three units. L* expresses the luminance and gives the relative brightness of the color ranging from total black (L* ¼ 0) to total white (L* ¼ 100).The terms a* and b* are coordinates of chromaticity, with a* representing the balance between green (negative values)and red (positive values) and b* representing the balance between blue (negative values) and yellow (positive values)

SECONDARY OUTCOMES:
Temperature | 3 month later
  Test tubes were equilibrated in water at 0◦C (cold) or 45-50 ◦C (warm) and applied for 5 s.
Light Touch | 3 month later
  The tactile sensation of the flap after surgery is assessed by Semmes-Weinstein monofilaments and the change in tactile sense is detected at least 3 months after surgery.
Two-point Discrimination（2PD） | 3 month later
  Two-point Discrimination of the flap after surgery was assessed by Touch-Test discriminator, and changes in 2PD were detected at least 3 months after surgery.
Flap Elasticity | 3 month later
  The elasticity of the flap after surgery was assessed by CK-MC960 and the change in elasticity was measured at least 3 months after surgery.
Melanin Content | 3 month later
  The melanin content of the flap after surgery was evaluated by Antera 3D, and the change of melanin was detected at least 3 months after surgery.
Hemoglobin Content | 3 month later
  The hemoglobin content of the flap after surgery was evaluated by Antera 3D, and the change of melanin was detected at least 3 months after surgery.
Satisfaction questionnaire | 3 month later
  At least 3 months after the patient's surgery, use a self-made satisfaction questionnaire to obtain patient satisfaction
Scar scaling | 6 month later
  The scar around the flap after surgery was evaluated by Patient and Observer Scar Assessment and the scar was assessed at least 6 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, the Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ensat F, Greindl M, Skreiner A, Schubert H, Hladik M, Stuflesser A, Spies M, Wechselberger G. Colorimetric examination of typical free flap donor sites and comparison to recipient sites in the extremities. J Reconstr Microsurg. 2013 Jan;29(1):21-6. doi: 10.1055/s-0032-1326734. Epub 2012 Oct 23. PMID 23093467
- [Result] Netscher D, Armenta AH, Meade RA, Alford EL. Sensory recovery of innervated and non-innervated radial forearm free flaps: functional implications. J Reconstr Microsurg. 2000 Apr;16(3):179-85. doi: 10.1055/s-2000-7549. PMID 10803620
- [Result] Ma X, Li Y, Li W, Liu C, Peng P, Song B, Xia W, Yi C, Lu K, Su Y. Reconstruction of Large Postburn Facial-Scalp Scars by Expanded Pedicled Deltopectoral Flap and Random Scalp Flap: Technique Improvements to Enlarge the Reconstructive Territory. J Craniofac Surg. 2017 Sep;28(6):1526-1530. doi: 10.1097/SCS.0000000000003902. PMID 28749842
- [Result] Ma X, Li Y, Li W, Liu C, Liu H, Xue P, Cui J. Reconstruction of Facial-Cervical Scars With Pedicled Expanded Deltopectoral Flap. J Craniofac Surg. 2017 Sep;28(6):1554-1558. doi: 10.1097/SCS.0000000000003901. PMID 28708657
- [Result] Abrar Y, Muntaha ST, Khan K, Hameed U. Successful Use of Deltopectoral Flap in Reconstruction of Defect Caused by Squamous Cell Carcinoma. J Coll Physicians Surg Pak. 2018 Jun;28(6):S125-S127. doi: 10.29271/jcpsp.2018.06.S125. PMID 29866245
- [Result] Ding J, Li Y, Li W, Liu C, Liu H, Cui J, Su Y, Ma X. Use of expanded deltopectoral skin flaps for facial reconstruction after sizeable benign tumor resections. Am J Transl Res. 2018 Jul 15;10(7):2158-2163. eCollection 2018. PMID 30093952
- [Result] Okochi M, Okochi H, Sakaba T, Ueda K. The Reconstruction of the Donor Site of DP Flap Using Thoracodorsal Artery Perforator Flap. Plast Reconstr Surg Glob Open. 2017 Oct 23;5(10):e1521. doi: 10.1097/GOX.0000000000001521. eCollection 2017 Oct. PMID 29184736
- [Result] Hwang K. The Origins of Deltopectoral Flaps and the Pectoralis Major Myocutaneous Flap. J Craniofac Surg. 2016 Oct;27(7):1845-1848. doi: 10.1097/SCS.0000000000003057. PMID 27763977
- [Result] Ibrahim A, Atiyeh B, Karami R, Adelman DM, Papazian NJ. The Deltopectoral Flap Revisited: The Internal Mammary Artery Perforator Flap. J Craniofac Surg. 2016 Mar;27(2):e189-92. doi: 10.1097/SCS.0000000000002445. PMID 26854779
- [Result] Murono S, Ishikawa E, Nakanishi Y, Endo K, Kondo S, Wakisaka N, Yoshizaki T. Closure of tracheoesophageal fistula with prefabricated deltopectoral flap. Asian J Surg. 2016 Oct;39(4):243-6. doi: 10.1016/j.asjsur.2014.01.003. Epub 2014 Mar 25. PMID 24674898
- [Result] Aldelaimi TN, Khalil AA. Reconstruction of Facial Defect Using Deltopectoral Flap. J Craniofac Surg. 2015 Nov;26(8):e786-8. doi: 10.1097/SCS.0000000000002056. PMID 26595007
- [Result] Moreno-Sanchez M, Gonzalez-Garcia R, Ruiz-Laza L, Manzano Solo de Zaldivar D, Moreno-Garcia C, Monje F. Closure of the Radial Forearm Free Flap Donor Site Using the Combined Local Triangular Full-Thickness Skin Graft. J Oral Maxillofac Surg. 2016 Jan;74(1):204-11. doi: 10.1016/j.joms.2015.08.003. Epub 2015 Aug 7. PMID 26342949
- [Result] Kesting MR, MacIver C, Wales CJ, Wolff KD, Nobis CP, Rohleder NH. Surface-optimized free flaps for complex facial defects after skin cancer. J Craniomaxillofac Surg. 2015 Nov;43(9):1792-7. doi: 10.1016/j.jcms.2015.08.010. Epub 2015 Aug 20. PMID 26355025
- [Result] Yangqun L, Yong T, Wen C, Zhe Y, Muxin Z, Lisi X, Chunmei H, Yuanyuan L, Ning M, Jun F, Weixin W. [Reconstruction of facial soft tissue defects with pedicled expanded flaps]. Zhonghua Zheng Xing Wai Ke Za Zhi. 2014 Sep;30(5):326-9. Chinese. PMID 25522480
- [Result] Beugels J, Cornelissen AJM, Spiegel AJ, Heuts EM, Piatkowski A, van der Hulst RRWJ, Tuinder SMH. Sensory recovery of the breast after innervated and non-innervated autologous breast reconstructions: A systematic review. J Plast Reconstr Aesthet Surg. 2017 Sep;70(9):1229-1241. doi: 10.1016/j.bjps.2017.05.001. Epub 2017 May 24. PMID 28687258
- [Result] Germann G, Rudolf KD, Levin SL, Hrabowski M. Fingertip and Thumb Tip Wounds: Changing Algorithms for Sensation, Aesthetics, and Function. J Hand Surg Am. 2017 Apr;42(4):274-284. doi: 10.1016/j.jhsa.2017.01.022. PMID 28372640
- [Result] Zhao G, Wang B, Zhang W, Tang P, Chen C. Sensory reconstruction in different regions of the digits: A review of 151 cases. Injury. 2016 Oct;47(10):2269-2275. doi: 10.1016/j.injury.2016.07.035. Epub 2016 Jul 27. PMID 27480911
- [Result] Cao G, Zheng D, Sun F, Shou K. [RECONSTRUCTION OF AVULSED INJURIES OF HEEL WITH A SENSORY PREFABRICATED FLAP]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2015 Feb;29(2):198-201. Chinese. PMID 26455150
- [Result] Xie A, Zhang J, Lu A, Yuan J, Wang B, Yang H, Zhang J, Wang H. [Effectiveness of retrograde island neurocutaneous flap pedicled with lateral antebrachial cutaneous nerve in treatment of hand defect]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2014 Dec;28(12):1498-501. Chinese. PMID 25826894
- [Result] Lu S, Chai Y. [Clinical application of sural fasciomyocutaneous perforator flap in repair of soft tissue defect in weight-bearing area of foot]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2014 Dec;28(12):1494-7. Chinese. PMID 25826893
- [Result] Trevatt AE, Filobbos G, Ul Haq A, Khan U. Long-term sensation in the medial plantar flap: a two-centre study. Foot Ankle Surg. 2014 Sep;20(3):166-9. doi: 10.1016/j.fas.2014.03.001. Epub 2014 Mar 18. PMID 25103702